CLINICAL TRIAL: NCT05852054
Title: Supporting Transitions to Primary Care Among Under-resourced, Postpartum Women: The STEP-UP Trial
Brief Title: Supporting Transitions to Primary Care Among Under-resourced, Postpartum Women (STEP-UP)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: AllianceChicago (Other); Cook County Health (Other Government)
Responsible Party: Principal Investigator, Stacy C Bailey, Associate Professor, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00217979
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes Mellitus; Hypertension in Pregnancy; Dysglycemia
MeSH Terms: conditions — Diabetes, Gestational; Hypertension, Pregnancy-Induced | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge, pragmatic design. Study sites deliver usual care until they are randomized to provide the STEP-UP intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients will receive the usual standard of care
- STEP-UP (Active Comparator): STEP-UP will promote linkage to primary care and ongoing chronic disease evaluation for postpartum women with prior GDM and/or HDP
  Interventions: Behavioral: OB Provider Clinical Decision Support (CDS); Behavioral: Patient Education (OB Visit); Behavioral: Text messaging; Behavioral: Patient Outreach; Behavioral: Primary Care Provider Clinical Decision Support (CDS); Behavioral: Patient Education (Primary Care Visit)

INTERVENTIONS:
Behavioral: OB Provider Clinical Decision Support (CDS) — When an eligible patients' chart is opened by a provider, the provider will be alerted to counsel patients about future risk for T2D and hypertension and the need to establish a primary care medical home. The alert will include a 'referral' to primary care and a brief guide with 'key points for counseling'. For patients with prior GDM, this will also include an option to order guideline-recommended oral glucose tolerance test (OGTT) with a single click.
  Arms: STEP-UP
Behavioral: Patient Education (OB Visit) — A 1-page document will be printed or delivered electronically for eligible patients after every postpartum OB visit during the STEP-UP condition. The document will encourage patients to know the risk and will describe the importance of routine primary care and chronic disease evaluation and management. It will also provide tips for lowering risk through lifestyle changes. Patient materials will be delivered in English or Spanish based on the structured EHR variable for preferred language.
  Arms: STEP-UP
Behavioral: Text messaging — At 3 months postpartum, all eligible patients who have not scheduled a primary care visit will receive a motivational text to prompt scheduling; a second text will be sent for those who still have not made an appointment. Among those who schedule a visit, a reminder text will be sent before the visit. Texts will be in English or Spanish based on patients' preferred language field in the EHR and written at a <5th grade reading level.
  Arms: STEP-UP
Behavioral: Patient Outreach — Patients who have not scheduled a primary care visit by 4 months postpartum will receive outreach from a trained coordinator who will assist with scheduling and help patients troubleshoot common barriers, such as concerns about transportation or cost.
  Arms: STEP-UP
Behavioral: Primary Care Provider Clinical Decision Support (CDS) — The CDS will notify the provider that the patient had a recent high-risk pregnancy and signal the need to counsel the individual about their future risk for T2D and/or hypertension and the need for ongoing care. A brief guide with 'key points for counseling' described in plain language will be provided. For patients with prior GDM, the CDS will also include an easy to access 'smartset' to order appropriate testing (A1c, FG, or OGTT) based on time since delivery and provider discussions with the patient.
  Arms: STEP-UP
Behavioral: Patient Education (Primary Care Visit) — A 1-page material will again be automatically printed or delivered electronically for eligible patients after their first primary care visit; it will replicate content from prior material provided after the OB visit.
  Arms: STEP-UP

SUMMARY:
STEP-UP will promote linkage to primary care and ongoing chronic disease evaluation for postpartum women with prior gestational diabetes mellitus (GDM) and/or hypertensive disorders of pregnancy (HDP).

DETAILED DESCRIPTION:
STEP-UP will promote linkage to primary care and ongoing chronic disease evaluation for postpartum women with prior gestational diabetes mellitus (GDM) and/or hypertensive disorders of pregnancy (HDP) by promoting:

1. counseling and referral to primary care, during OB visits, via electronic health record (EHR)-based clinical decision support (CDS)
2. dysglycemia testing for women with prior GDM, prompted via CDS during both OB and primary care visits
3. dissemination of understandable information on future risk and the need for ongoing evaluation generated automatically via the EHR and printed for patients with after-visit summaries (AVS)
4. motivational messaging and reminders supporting transitions of care delivered directly to patients via short message service (SMS) text messages
5. individualized outreach and support for those who need additional help arranging a primary care visit

We will utilize a stepped wedge design to achieve the study's specific aims, which are to:

Aim 1 Test the effectiveness of STEP-UP, compared with usual care, to improve patient: 1) knowledge of reproductive risks associated with T2DM and recommended self-care activities; 2) engage in self-care behaviors, including diet, physical activity, adherence to diabetes medications, and use of folic acid and most or moderately effective contraception, when indicated; and 3) clinical measures, including hemoglobin A1c, blood pressure, and LDL cholesterol.

Aim 2 Investigate the heterogeneity of STEP-UP intervention effects by patients' race, ethnicity, and language.

Aim 3 Assess the reach, adoption, implementation, maintenance and costs of STEP-UP components.

ELIGIBILITY:
Inclusion Criteria:

* Delivered during an accrual period,
* Had a chart diagnosis during their index pregnancy of GDM and/or HDP,
* Attended at least 1 prenatal care visit at a study site in the 6 months prior to delivery,
* Speak English or Spanish,
* Age 18 or older

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All trial participants will be women with gestational diabetes and/or hypertensive disorders of pregnancy; they will be accrued into the study upon delivery.
Enrollment: 1500 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Primary care visit (PCV) completion | 6 months
  Assess completion of a primary care visit (yes/no) within 6 months of delivery. Using procedures from a pilot study, the investigator will consider an encounter a PCV if it occurred by 6 months after the delivery date; had an assigned provider type of "nurse practitioner," "physician," "internal medicine," "family medicine," and/or "physician assistant;" and did not have an assigned provider type of "OB/GYN" and/or "certified nurse midwife." The PCV rate across STEP-UP vs. UC will be calculated by dividing eligible patients with greater than or equal to 1 PCV (numerator) by the denominator of all eligible patients.

SECONDARY OUTCOMES:
Completion of dysglycemia testing | 6 months
  Assess rates of testing for dysglycemia among eligible women who had a diagnosis of GDM in their index pregnancy. This binary outcome (yes/no) will be ascertained by the presence of a value from any dysglycemia test (e.g. A1c, fasting glucose, oral glucose tolerance test) at any time within the 6-month follow-up period. The testing rate across STEP-UP vs. UC will be calculated by dividing this numerator by the denominator of all eligible patients with GDM in their index pregnancy.
Orders for dysglycemia testing | 6 months
  Assess whether eligible patients have an order for any dysglycemia test (e.g. A1c, fasting glucose, oral glucose tolerance test) at any time during the 6-month follow-up period. This dichotomous outcome largely assesses the effectiveness of the provider-facing STEP-UP components. The investigator ascertain orders in this same way across STEP-UP and UC conditions. As an exploratory outcome, the investigator will examine the proportion of total tests ordered through the CDS versus the routine lab order entry mechanism. The investigator will also examine the association of orders with patient characteristics (e.g. age, BMI, race, ethnicity, language) and provider characteristics available in the EHR (i.e. physician vs. advanced practice provider, patient panel size).
Dysglycemia and hypertension cases detected | 6 months
  Assess the rate of dysglycemia and hypertension cases detected among eligible patients. Rate of detection for dysglycemia will be determined by the proportion of eligible patients with a prior diagnosis of GDM (i.e. denominator) who have a test value indicating dysglycemia according to ADA guidelines during follow-up (i.e. numerator). The rate of dysglycemia cases detected will be compared between STEP-UP and UC conditions. The investigator will run similar analyses for hypertension, using 2017 American College of Cardiology/American Heart Association criteria (hypertension: systolic blood pressure (SBP) greater than or equal to 130 mmHg or diastolic blood pressure (DBP)greater than or equal to 80 mmHg; stage 2 hypertension defined as SBP greater than or equal to 140 mmHg or DBP greater than or equal to 90 mmHg).

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Bailey, PhD MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Cook County Health, Chicago, Illinois
  - AllianceChicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT05852054/ICF_000.pdf